CLINICAL TRIAL: NCT00322309
Title: The Efficacy of Mirtazapine in Depressed Cocaine Dependent Subjects
Brief Title: Efficacy of Mirtazapine in Depressed Cocaine Dependent Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-22530
Record Dates: First submitted 2006-05-03; First posted 2006-05-05 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Cocaine Dependence; Depression
Keywords: Cocaine; Substance Abuse
MeSH Terms: conditions — Cocaine-Related Disorders; Depression; Substance-Related Disorders | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mirtazapine (Experimental): Mirtazapine administration as follows:
  Days 1-4 15mg of mirtazapine daily Days 5-9 30mg of mirtazapine daily Days 10-78 45mg of mirtazapine daily Days 79-81 30mg of mirtazapine daily Days 82-84 15mg of mirtazapine daily
  Interventions: Drug: Mirtazapine
- Placebo- Sugar pill (Placebo Comparator): Matched Placebo given daily days 1-84
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Placebo for days 1-4 Placebo for days 5-9 Placebo for days10-78 Placebo for days 79-81 Placebo for days 82-84
  Arms: Placebo- Sugar pill
Drug: Mirtazapine — Days 1-4 15mg Days 5-9 30 mg Days 10-78 45mg Days 79-81 30mg Days 82-84 15mg
  Other Names: Remeron
  Arms: Mirtazapine

SUMMARY:
This research study is being done to look at the safety of the medication Mirtazapine (Remeron) in people who have cocaine dependence and depression. Hypotheses I. Cocaine usage will be less in the mirtazapine treatment group (MG) than in the control group (CG). II. A greater increase in Clinician Global Impression (CGI) score will be observed in the MG than in the CG. Secondary Hypotheses: I. A greater decrease in Hamilton Rating Scale for Depression (HAM-D) and Hamilton Rating Scale for Anxiety (HAM-A) scores will be observed in the MG than in the CG. II. A greater decrease in HIV risk behaviors will be observed in the MG than in the CG. III. A greater improvement in sleep structure will be observed in the MG than in the CG. IV. The proportion of subjects experiencing severe adverse drug reactions that necessitate termination from the study by one of the study clinicians will not differ between the MG and CG. V. Retention will be greater in MG than in CG.

DETAILED DESCRIPTION:
Cocaine dependence is a significant public health problem associated with serious medical, psychiatric, social and economic consequences. It is generally accepted that the euphoria associated with cocaine use is a result of its action on reward pathways via antagonist properties at the dopamine transporter site; cocaine also inhibits reuptake of serotonin and norepinephrine. These actions are thought to underlie cocaine's potent reinforcing properties. With prolonged use, cocaine may deplete these neurotransmitters, affect postsynaptic receptor density, and elicit an overall dysregulation of these neurotransmitter systems. These longer term consequences may account for the post-cocaine depressive symptoms often claimed by cocaine users to contribute to relapse. Treatment for cocaine dependence at the present is primarily psychosocial/behavioral. Currently there is no pharmacological agent approved for treatment of cocaine dependence in conjunction with psychosocial interventions. Several drugs currently approved for other indications are presently under consideration for treatment of cocaine dependence based on their known mechanisms and sites of action. Current approaches include strategies to (1) block the effects of cocaine, (2) substitutes for cocaine, (3) reduce craving or enhance the addict's ability to manage his/her response to craving, and (4) treat underlying conditions (or consequences of cocaine use) that may predispose toward dependence.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnosis of cocaine dependence.
* HAM-D score of 12 or above and history of autonomous depression, defined as meeting DSM-IV criteria for major depression or dysthymic disorder during any lifetime period of abstinence of 30 days or longer.
* At least one urine toxicology positive for cocaine benzoylecgonine (BE) over the consecutive two-week baseline screening period during which 6 urine samples have been obtained
* Males and non-pregnant, non-nursing females, 18-64 years of age (inclusive).
* Individuals able to give written informed consent and willing to comply with all study procedures.

Exclusion Criteria:

* Any Axis I diagnosis that, in the opinion of the Principal Investigator, may interfere with the course of the trial.
* Physiological dependence on alcohol or opiates requiring medical detoxification.
* A medical or neurological illness that in the clinical judgment of the investigator would make study compliance difficult or contraindicate the use of mirtazapine.
* Any clinically significant abnormal lab values or liver function tests (LFTs) which are greater than 3 times the normal limit.
* The need or intention to use concurrently with or within four weeks prior to study drug administration, any of the following medications: monoamine oxidase inhibitors and/or sibutramine. In addition, other medications such as alpha2-agonists and medications which affect the enzymes Cytochrome P450 1A2 (CYP1A2), Cytochrome P450 2D6 (CYP2D6), Cytochrome P450 3A4 (CYP3A4) (as inhibitors, substrates, or inducers), and serotonin modulators should be used with caution. The research physician will decide on this issue. A listing of these substances may be found in Appendix I.
* Females of childbearing potential who do NOT agree to use a medically acceptable method of birth control (barrier, intrauterine device (IUD), oral or depot contraceptive medication, or complete abstinence).
* Positive pregnancy test.
* Breastfeeding
* Known drug allergy or sensitivity to mirtazapine.
* Participation in an investigational drug or device study within 1 month of enrollment in the present study.
* Enrollment in an opiate-substitution (i.e., methadone, levo acetyl methadol (LAAM)) treatment program within 45 days of enrolling in the present study.
* Individuals having taken LAAM, methadone or naltrexone within 14 days of enrollment in the present study.
* Individuals who, in the clinical judgment of the Investigator, are actively and acutely suicidal.
* Subjects, who in the opinion of the investigator, have a medical condition that may interfere with study assessments and/or put them at undue risk.
* Subjects, who in the opinion of the investigator, will have difficulty complying with study procedures.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-09; Primary Completion 2009-07 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Afshar, MD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at the Boston University Psychiatry Associates Clinical Studies Unit
Groups:
- Mirtazapine: Mirtazapine daily:
  Days 1-4 15mg Days 5-9 30mg Days 10-78 45mg Days 79-81 30mg Days 82-84 15mg
- Placebo: Matched placebo given daily days 1-84
Period: Overall Study
Arm/Group | Mirtazapine | Placebo
Started | 11 | 13
Completed | 9 | 9
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Subjects received matched placebo capsules
- Total: Total of all reporting groups
Arm/Group | Mirtazapine | Placebo | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 13 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (5.6) | 47.2 (6.7) | 45.7 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 11 | 13 | 24
Ln Urine Benzoylecgonine Conc [Mean (Standard Deviation); unit: ln (ng/ml)] — Baseline urine LB BE concentrations were obtained during the screening sessions.
  ln (ng/ml) | 9.3 (1.7) | 9.1 (2.4) | 9.2 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Ln Benzoylecgonine Concentration
Time Frame: Week 11
Population: Data was analyzed for all subjects who provided data for the second assessment visit.
Measure: Mean (Standard Deviation); unit: ln (ng/ml)
Arm/Group | Mirtazapine | Placebo
Number analyzed (Participants) | 11 | 13
ln (ng/ml) | 9.8 (1.8) | 7.9 (3.2)
Statistical Analysis 1: Comparison: Mirtazapine vs Placebo; It was hypothesized that there would be no significant difference between the two treatment groups for benzoylecgonine data collected for Week 11; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = 1.9, Standard Deviation 2.6

2. Secondary Outcome: The Clinical Global Impression Observer (CGI-O)Comparison for Week 11
Description: Clinician's overall assessment of the subjects global functioning including the severity of the subject's cocaine use, cocaine seeking, use of other drugs, psychiatric symptoms, medical problems, maladaptive family/social coping, and coping with issues related to employment, housing, and legal issues. Totals range between 7 (for none) to 56 for most severe.
Time Frame: Week 11
Population: Data was analyzed fof all subjects for whom data from the second evaluation visit was available
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mirtazapine | Placebo
Number analyzed (Participants) | 11 | 13
Scores on a scale | 29.9 (4.8) | 23.1 (8.5)
Statistical Analysis 1: Comparison: Mirtazapine vs Placebo; It was hypothesized that means scores for the CGI-O would not differ significantly for these values obtained in the final treatment week, Week 11; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = 6.8, Standard Deviation 6.6

3. Secondary Outcome: Hamilton Depression Rating Scale
Description: Subjects are assessed on 24 characteristics of depressive disorders. Scale scores may range from 0 for no depressive symptoms to 75.
Time Frame: Week 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Mirtazepine: Mirtazapine daily:
  Days 1-4 15mg Days 5-9 30mg Days 10-78 45mg Days 79-81 30mg Days 82-84 15mg
- Placebo: Matched placebo capsules
Arm/Group | Mirtazepine | Placebo
Number analyzed (Participants) | 11 | 13
Scores on a scale | 7.2 (4.7) | 6.7 (6.1)
Statistical Analysis 1: Comparison: Mirtazepine vs Placebo; It hypothesized that the two treatment groups would not differ significantly with respect to the total HAM-D scores obtained in the final week of the study (Week 11); Test type: Superiority or Other; p > 0.05, t-test, 2 sided — This analysis involves a between group comparison; Mean Difference (Final Values) = 0.05, Standard Deviation 5.4

4. Secondary Outcome: Pill Count
Description: Percentage of medication capsules administered based on the ratio of the number of capsules administered to the total number dispensed for entire period during which subjects were in treatment.
Time Frame: Weeks 1 to 11
Measure: Mean (Standard Deviation); unit: Percentage of dispensed capsules
Arm/Group | Mirtazapine | Placebo
Number analyzed (Participants) | 11 | 13
Percentage of dispensed capsules | 91 (21) | 91 (15)
Statistical Analysis 1: Comparison: Mirtazapine vs Placebo; It was hypothesized that there would be no significant difference in the mean percentage of capsules of those dispensed between the two groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Percent of capsules administered does not differ significantly between the two groups; Mean Difference (Net) = 0, Standard Deviation 18

5. Secondary Outcome: Percent Urines Positive for Riboflavin
Description: This measure of adherence was determined by finding the percent of total urines examined that were positive for riboflavin, which had been added to each medication tablet.
Time Frame: Weeks 1-11
Measure: Mean (Standard Deviation); unit: Percentage of total urines examined
Arm/Group | Mirtazapine | Placebo
Number analyzed (Participants) | 11 | 13
Percentage of total urines examined | 93.5 (7.6) | 93.5 (9.5)
Statistical Analysis 1: Comparison: Mirtazapine vs Placebo; It was hypothesized that there would not be a significant difference between the two groups in the mean percent of urines positive for riboflavin; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; Mean Difference (Net) = 0, Standard Deviation 8.5

ADVERSE EVENTS:
Groups:
- Mirtazapine Daily: Days 1-4 15mg Days 5-9 30mg Mirtazapine: Mirtazapine daily:
  Days 1-4 15mg Days 5-9 30mg Days 10-78 45mg Days 79-81 30mg Days 82-84 15mg
- Placebo: Matched placebo
Arm/Group | Mirtazapine Daily: Days 1-4 15mg Days 5-9 30mg Mirtazapine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 2/11 | 1/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirtazapine Daily: Days 1-4 15mg Days 5-9 30mg Mirtazapine (N=11) | Placebo (N=13)
Sleepiness (Nervous system disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mood Swings (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Fainting (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes